CLINICAL TRIAL: NCT02390635
Title: PET/MR, PET/CT and Whole Body MR in Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: PET/MRI, 18F-FDG PET/CT and Whole Body MRI in Finding Extramedullary Myeloid Leukemia in Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0616; NCI-2015-00525 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0616 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Acute Promyelocytic Leukemia With PML-RARA
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute | interventions — Fluorodeoxyglucose F18; Gadolinium; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (18F-FDG PET/CT, whole body PET/MRI) (Experimental): Patients receive gadolinium IV and undergo whole body PET/MRI comprising diffusion weighted imaging and 3D FSPGR-DE with and without fiducial markers. Patients then undergo 18F-FDG PET/CT before start treatment for acute myeloid leukemia.
  Interventions: Procedure: Computed Tomography; Procedure: Diffusion Weighted Imaging; Radiation: Fludeoxyglucose F-18; Drug: Gadolinium; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Three-Dimensional Spoiled Gradient MRI

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 18F-FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Diffusion Weighted Imaging — Undergo whole body PET/MRI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DW-MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Radiation: Fludeoxyglucose F-18 — Undergo 18F-FDG PET/CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Gadolinium — Given IV
  Other Names: Gd
Procedure: Magnetic Resonance Imaging — Undergo whole body PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo 18F-FDG PET/CT and whole body PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Three-Dimensional Spoiled Gradient MRI — Undergo whole body PET/MRI
  Other Names: 3-Dimensional Fast Spoiled Gradient; 3D Fast Spoiled Gradient Recalled MRI; 3D FSPGR; 3DFSPGR; FSPGR; FSPGR MRI; SPGR; SPGR MRI; Three-Dimensional Spoiled Gradient-Echo MR

SUMMARY:
This pilot phase I trial studies how well positron emission tomography (PET)/magnetic resonance imaging (MRI), fludeoxyglucose F-18 (18F-FDG) PET/computed tomography (CT), and whole body MRI work in finding extramedullary myeloid leukemia in patients with newly diagnosed acute myeloid leukemia. Extramedullary myeloid leukemia is a type of cancer found outside of the bone marrow and can be hard to detect with routine bone marrow monitoring, such as bone marrow aspirations. Diagnostic procedures, such as PET/MRI, 18F-FDG PET/CT and whole body MRI, may help find and diagnose extramedullary myeloid leukemia in patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the incidence of extramedullary myeloid leukemia (EML) in patients with newly diagnosed acute myeloid leukemia (AML), including acute promyelocytic leukemia (APL), by imaging criteria using PET/MR (magnetic resonance), whole body MR, and PET/CT.

SECONDARY OBJECTIVES:

I. To qualitatively and quantitatively assess PET/MR and PET/CR that will be performed with and without fiducial markers, and to correlate these findings with clinical outcomes of treatment response, relapse, and patterns of relapse.

II. Correlate findings of EML as in the primary objectives with clinical outcomes of treatment response, relapse, and patterns of relapse including location of relapse compared to site of EML.

OUTLINE:

Patients receive gadolinium intravenously (IV) and undergo whole body PET/MRI comprising diffusion weighted imaging and 3-dimentional (3D) fast spoiled gradient echo dual echo (FSPGR-DE) with and without fiducial markers. Patients then undergo 18F-FDG PET/CT before start treatment for acute myeloid leukemia.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML
* Non-English speaking subjects will be included. Verbal Translation Preparative Sheet (VTPS) short form will be utilized in consenting non-English speaking subjects.

Exclusion Criteria:

* Patients with contraindications to MR
* Patients with a known allergy to MR contrast agents
* Uncontrollable claustrophobia
* Recipients of more than minimal anti-leukemia treatment, with minimal treatment defined as: leukapheresis, hydroxyurea, or Cytarabine more than 1 g per square meter.
* Patients with secondary or relapsed AML or APL should be excluded.
* Patients with known extramedullary leukemia
* Positive pregnancy test in a female of childbearing potential
* Younger than 18 years
* Greater than 400 pounds in weight
* Patients with uncontrolled diabetes
* Cognitive impaired adults or prisoners will be excluded
* Estimated glomerular filtration rate (eGFR <30) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of extramedullary myeloid leukemia (EML) | At time of imaging
  Defined as increased fludeoxyglucose F-18 uptake on positron emission tomography (PET)/computed tomography and increased signal on T2 weighted imaging or diffusion weighted imaging and enhancement in soft tissue on whole body PET/magnetic resonance imaging. Estimates and 95% confidence intervals for the incidence of EML will be reported for each imaging modality based on the exact Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Dawid Schellingerhout, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org